CLINICAL TRIAL: NCT06149182
Title: Does the First Interview Matter: A Randomized Trial Comparing Life Stress Interview Versus a Standard Psychiatric Intake Interview for Patients With Functional Somatic Disorder
Brief Title: Does the First Interview Matter: A Comparing Life Stress Interview Versus a Standard Psychiatric Intake Interview for Patients With Functional Somatic Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Maroti (Other)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor-Investigator, Daniel Maroti, Researcher, Med.dr, Stockholm University
Organization: Stockholm University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: StockholmU
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Functional Somatic Disorder; Somatic Symptom Disorder
Keywords: Functional somatic disorder; Somatic symptom disorder; life stress interview; emotional awareness and expression therapy; intensive short term psychodynamic therapy; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life stress interview/therapeutic interview (Experimental): Revised "Life stress interview" according to protocol from emotional awareness and expression therapy
  Interventions: Behavioral: Life stress interview according to EAET
- Psychiatric interview (Active Comparator): Psychiatric interview (M.I.N.I. etc) according to "Region stockholm - basutredning"
  Interventions: Behavioral: Psychiatric interview according to "region stockholm - basutredning"

INTERVENTIONS:
Behavioral: Life stress interview according to EAET — This interview has the aim to jointly explore potential emotional factors contributing to patients functional somatic symptoms. While exploring this, it has the aim to not only describe such potential patterns but also emotionally process them.
  Arms: Life stress interview/therapeutic interview
Behavioral: Psychiatric interview according to "region stockholm - basutredning" — This interview has the aim to gain enough information to diagnose some of the main psychiatric disorders
  Arms: Psychiatric interview

SUMMARY:
Functional somatic syndromes (e.g. irritable bowel syndrome, fibromyalgia) and medically unexplained symptoms (e.g. chronic primary pain) are very common in primary care. These patients make 14 times more doctor visits than the general population, but describe themselves as less satisfied with the care they receive. Although Region Stockholm in Sweden recently developed care flows based on 'step up' care for the most common patient groups in primary care, patients with functional or medically unexplained symptoms are not mentioned.

Short-term psychodynamic therapies such as Emotional Awareness and Expression Therapy (EAET) and Intensive Short Term Psychodynamic Therapy (ISTDP) have recently been evaluated in three systematic reviews and show good results for patients with medically unexplained symptoms. Short-term psychodynamic therapy considers that good treatment outcomes for patients with functional somatic syndromes can be achieved by increasing awareness of emotions and teaching patients to better experience, express and regulate emotions. In several randomized studies, short-term psychodynamic therapy has shown good effects even compared to other treatments, including cognitive behavioral therapy (CBT).

The overall purpose of this research project is to to evaluate psychodynamic emotion-focused interventions (EAET and ISTDP) for patients with medically unexplained symptoms and high health care consumption. The project includes several studies that will clarify effects and contribute to information on how care flows in primary care for the patient group can be created.

The research question for this specific study is:

Can a therapeutic interview (so-called "EAET life-stress interview") focusing on emotional factors in comparison to a psychiatric interview (so-called "basic assessment") contribute to increased interest in psychological treatment and reduction of physical and psychiatric symptoms in patients with medically unexplained symptoms with relatively high health care consumption? Does the order of interview interventions matter?

ELIGIBILITY:
Inclusion Criteria:

1. The research subject certifies that he/she has undergone medical assessment for his/her physical symptoms.
2. The subject must have visited a physician at least three times in the last year.
3. The subject rates either moderate distress from bodily symptoms in the PHQ-15 (over 10 points) or severe distress from a single bodily symptom (at least 2 points for this symptom).
4. The research participants expresses interest in investigating whether emotional factors such as stress may contribute to symptoms.
5. Research subjects either affirm the presence of emotionally difficult life events (affirm at least 1 such event in the ACE-10 or reach the proposed cut-off point of 21p in the PCL-5).
6. Drugs used should have been stable for at least 1 month.

Exclusion Criteria:

1. Research subjects suffer from ongoing substance abuse (alcohol or drugs) or are deemed to have serious mental illness (psychotic illness, suicidal ideation, antisocial personality disorder etc).
2. The research subjects have ongoing medication of a clearly addictive and sedative nature (e.g. benzodiazipines).
3. The research subject participates in other psychological treatment focusing on physical symptoms. However, other psychological treatment is allowed where the support therapy does not take place more often than once a month.
4. The research subject does not master the Swedish language sufficiently to be able to assimilate written material in Swedish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scales according to EURONET-SOMA | Change from pre to follow up (6 weeks after interview)
  Visual analogue scale 0-10 for symptom intensity and symptom interference. Higher scores indicates worse symptom/functioning.
PHQ-15 | Change from pre to follow up (6 weeks after interview)
  Ratings 0-2 on how troublesome somatic symptoms are experienced. Higher scores indicates worse symptom/functioning.

SECONDARY OUTCOMES:
Numeric Rating Scales according to EURONET-SOMA | Change from pre to post (within 1 week after interview)
  Visual analogue scale 0-10 for symptom intensity and symptom interference. Higher scores indicates worse symptom/functioning.
PHQ-15 | Change from pre to post (within 1 week after interview)
  Ratings 0-2 on how troublesome somatic symptoms are experienced. Higher scores indicates worse symptom/functioning.
PHQ-9 | Change from pre to post (within 1 week after interview) and follow up (6 weeks after interview)
  Ratings 0-3 on impact of depressive symptoms. Higher scores indicates worse symptom/functioning.
GAD-7 | Change from pre to post (within 1 week after interview) and follow up (6 weeks after interview)
  Ratings 0-3 on impact of anxiety symptoms.Higher scores indicates worse symptom/functioning.
PCL-5 | Change from pre to post (within 1 week after interview) and follow up (6 weeks after interview)
  Ratings 0-4 on impact of post traumatic symptoms. Higher scores indicates worse symptom/functioning.
DERS-16 | Change from pre to post (within 1 week after interview) and follow up (6 weeks after interview)
  Ratings on emotional (dys)regulation. Higher scores indicates worse symptom/functioning.
Sheehan Disability Scale (SDS) | Change from pre to post (within 1 week after interview) and follow up (6 weeks after interview)
  Visual analogue scale 0-10 for symptom interference in daily life. Higher scores indicates worse symptom/functioning.
IPQ-R | Change from pre to post (within 1 week after interview) and follow up (6 weeks after interview)
  Ratings on illness beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lilliengren, PhD, Principal Investigator — Stockholm University
Locations (1):
- Stockholm University, Stockholm, Sweden